CLINICAL TRIAL: NCT04532242
Title: Investigating the Neural Systems That Support the Reappraisal Tactics Leading to Positive Emotion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Denver (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Principal Investigator, Kateri McRae, Professor, University of Denver
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1606445-A
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Behavior
Keywords: cognitive reappraisal; cognition
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI Participants (Experimental): Participants will be scanned in an fMRI session lasting approximately 45-50 minutes and will be shown negative images for which they will have to take on a cognitive reappraisal tactic. All participants will be taken through the scanner with the same reappraisal protocol for each participant.
  Interventions: Behavioral: Cognitive reappraisal

INTERVENTIONS:
Behavioral: Cognitive reappraisal — Participants will be trained to follow instructions to look/respond naturally or use cognitive reappraisal to reframe or reconsider a negative picture to decrease negative emotion.

SUMMARY:
Community participants will visit the neuroimaging facilities at CU Boulder for a single experimental session. In all studies, participants will complete pre-task questionnaires (trait measures), and a brief mood measure, followed by a task training in which a research assistant describes and gives examples of cognitive reappraisal in response to negative images. Then, participants complete an event-related, picture-based cognitive reappraisal task for 30-45 minutes, during which whole-brain BOLD signal will be collected. Following the task, participants will once again respond to a mood measure, and answer a series of questions regarding the task they have completed, including difficulty of regulation, or any images that were personally relevant.

The researchers predict that the positive emotion induction will result in powerful effects on self-reported emotion which may or may not interact with the cognitive reappraisal condition. Participants will be trained to use reappraisal to increase positive emotion, and they will be asked to respond with the reappraisal tactic category that best fits the reappraisal they used for each image. The researchers predict greater use of future-focused tactics will be associated with greater reappraisal success, which in turn will result in greater recruitment of vmPFC and connectivity between vmPFC and other prefrontal regions.

DETAILED DESCRIPTION:
For all studies, participants will be recruited via paper and electronic flyers on campus and in the surrounding communities. Interested participants will be screened via phone, email and/or web form to assess eligibility according to criteria listed elsewhere. Should participants qualify, they will be invited to complete a single laboratory session at the Intermountain Neuroimaging Facility at CU Boulder. Participants will be sent a copy of the consent form to read in advance of their visit, and to keep for their records.

Once arriving at the laboratory, participants will complete the consent process, in which a research assistant trained in ethical principles regarding human subjects research will answer any questions about the consent form and verbally reinforce the key rights of the participants outlined there. Once both parties are satisfied, consent forms will be signed.

Participants will then complete a mandatory day-of MRI eligibility form to ensure scanner compatibility has not changed since the initial screening (done by phone, email or webform). Females who are unable to indicate "no" to the question, "is it possible that you are pregnant?" will be asked to take a pregnancy test provided at the MR facility. Participants will change into MRI- compatible clothes or scrubs. Participants will sit with a trained research assistant/experimenter who will give an overview of the entire session, and then begin training for the cognitive reappraisal task. This training takes 10-15 minutes. During the training, the experimenter will offer several possible reappraisals of negative images and allow the participants to offer their own as well, providing encouragement and feedback. During this training, the experimenter will also go over the method of encouragement and feedback. During this training, the experimenter will also go over the method of responding (using an external button box). Participants will be reminded during training that they may stop the experiment at any point if the pictures are too upsetting.

Immediately following task training, participants will make a general mood rating using the PANAS. Then, participants will be screened one final time for metal in or near their bodies at the door to the shielded MRI room, then be placed in the MRI scanner by a certified, full-time MRI technician. Participants will be reminded they can stop the experiment at any point if they are physically uncomfortable or become claustrophobic, and will be outfitted with a panic button to indicate that they wish to stop the experiment immediately once it has begun. After the initial structural and calibration scans, participants will complete the reappraisal task. The task will take 40-50 minutes (broken up into 4-5 separate functional runs in the scanner, with each run taking around 10 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Community members ages 18-55
* Fluent in English
* Without present psychotic symptoms

Exclusion Criteria:

* None

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported emotion ratings | During the task intervention which will last 50 minutes
  Participants will be rating their negative and positive emotions during the intervention. They will be asked "How positive do you feel?" and "How negative do you feel?" after each image and will answer on a scale of 1-9 with 1 being low ("I don't feel positive at all" or "I don't feel negative at all") to 9 ("I feel very positive" or "I feel very negative").
Whole brain BOLD signal | Immediately after the intervention
  Changes in blood oxygen dependent level (EPI sequences) from the whole brain collected in a 3T MRI scanner with a head-coil specifically for fMRI.

SECONDARY OUTCOMES:
Mood ratings | Pre-intervention and immediately after the intervention
  Pre- and post-task mood as measured by the Positive and Negative Affect Schedule (PANAS) will be taken before and after the intervention. The PANAS is a 20-question questionnaire rated on a scale of 1 to 5 (with 1 being "very slight or not at all" and 5 being "extremely"). Questions 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19 represent the positive affect scale with scores ranging between 10 and 50 (the higher the score, the higher the levels of positive affect). Questions 2, 4, 6, 7, 8, 11, 13, 15,18, and 20 represent the negative affect scale with scores falling between 10 and 50 (lower scores represent lower levels of negative affect).
Task difficulty | Immediately after the intervention
  The next batch of questions will ask the participant questions about the difficulty of the task. An example question is "How difficult was it to follow the 'LOOK' instruction?" Participants will be rating the level of difficulty on a scale of 1 to 7 with 1 being "not difficult at all" to 7 being "very difficult".
Task compliance | Immediately after intervention
  Participants will be asked about self-reported task compliance. For example, one question will ask "What percentage of the time were you able to follow the "LOOK" instruction?" The participants will be rating their self-compliance for each task from 0% (non-compliant) to 100% (fully compliant).
Experience with task images | Immediately after intervention
  Participants will be asked whether they have any experience with reappraisal or the specific images presented in the task. The first question will ask "Have you ever been trained to change your emotions by changing the way you think (in therapy, or in another experiment, or anywhere else)?" Participants can choose "Yes" or "No" for this question. The participant will have to extrapolate if they have changed their emotions before using a fill in the blank. The next question will ask "Have you ever seen any of these exact emotional images before?" The participant then once again will be asked to extrapolate which images they have seen and what emotional response was generated by these images using a fill in the blank option.

OTHER OUTCOMES:
Depression trait differences | Baseline
  The participants will be given the Beck's Depression Inventory(BDI-II) which measures symptoms of depression and will be used to examine any between-subjects trait differences. The BDI-II is a 21 self-report measure looking at symptoms of depression with ratings falling between 0 and 3 (0 being "not at all" and 3 would indicate experiencing these symptoms on a constant basis).
Emotional regulation trait differences | Baseline
  The Emotion Regulation Questionnaire (ERQ) looks at methods of regulating emotions and will be used to examine any between-subjects trait differences. The ERQ is a 10-item self-report questionnaire assessing the use of two strategies to alter emotions: cognitive reappraisal and expressive suppression. The scale is rated on a 7-point Likert scale with 1 being "strongly disagree" and 7 being "strongly agree". Six items are categorized as using cognitive reappraisal while four of the items assess expressive suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Kateri McRae, Ph.D., Principal Investigator — University of Denver
Locations (1):
- University of Denver, Denver, Colorado, United States